CLINICAL TRIAL: NCT01561378
Title: Intranasal Insulin for Neuroprotection in Elderly Cardiac Surgery Patients
Brief Title: Cardiac Surgery Neuroprotection Study in Elders
Acronym: CNS-Elders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2010-538; R03AG040673 (NIH)
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Post-operative Cognitive Decline; Post-operative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Insulin Aspart; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin (Experimental): Aspart Insulin 40 IU intranasal spray via intranasal mucosal atomizer device, four times a day for 7 days or until hospital discharge, whichever occurs first
  Interventions: Drug: Aspart insulin; Device: Intranasal mucosal atomizer device
- Normal saline (Placebo Comparator): Normal saline (0.9% sodium chloride solution) intranasal spray via intranasal mucosal atomizer device, four times a day for 7 days or until hospital discharge, whichever occurs first
  Interventions: Drug: Normal saline; Device: Intranasal mucosal atomizer device

INTERVENTIONS:
Drug: Aspart insulin — 40 IU of aspart insulin (200 microliters per nostril) will be administered intranasally using an intranasal mucosal atomizer device within 2 hours prior to surgery, and then four times a day for 7 days or until hospital discharge (whichever occurs first)
  Other Names: NovoLog
  Arms: Insulin
Drug: Normal saline — 200 microliters of normal saline will be administered per nostril using an intranasal mucosal atomizer device within 2 hours prior to surgery, and then four times a day for 7 days or until hospital discharge (whichever occurs first)
  Other Names: 0.9% sodium chloride solution
  Arms: Normal saline
Device: Intranasal mucosal atomizer device — Insulin and placebo will be drawn into identical syringes. Nurses will administer the insulin or placebo by connecting the mucosal atomizer device (MAD) to the syringe, placing the MAD tip in the nostril and compressing the syringe plunger to spray atomized solution into the nasal cavity.
  Other Names: mucosal atomizer device, MAD

SUMMARY:
The goal of this study is to determine the potential ability of intranasal insulin to prevent post-operative cognitive decline and post-operative delirium in an elderly cardiac surgery population.

DETAILED DESCRIPTION:
Nearly half of all intensive care unit (ICU) admissions consist of adults > 65 years old, an age group that is at high risk for developing cognitive decline and delirium in the ICU. Over 50% and 70% of critically ill cardiac surgery patients develop post-operative delirium (POD) and post-operative cognitive decline (POCD), respectively. These two forms of acute cognitive dysfunction are associated with increased mortality and poor functional recovery. While distinct conditions, POD has been associated with the subsequent development of POCD, suggesting a mechanistic link.

No proven pharmacologic treatments targeting the prevention of both POD and POCD in elderly patients exist to date. Recent data suggest that insulin administered into the central nervous system via intranasal delivery improves cognitive function in elderly patients with Alzheimer's disease and mild cognitive impairment. However, its utility in preventing POD and POCD in elderly critically ill patients has not been investigated.

The hypothesis of this study is that intranasal insulin can prevent POD and POCD in elderly critically ill patients admitted to the intensive care unit after undergoing cardiac surgery. To test this hypothesis, this randomized, placebo-controlled, double-blinded Phase II study will enroll 60 patients >= 65 years old undergoing elective coronary artery bypass graft and/or valve surgery requiring cardiopulmonary bypass, and will treat them with either 40 IU of aspart insulin or placebo intranasally before surgery and then four times a day for 7 days or until hospital discharge (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. elderly patients (>=65 years old)
2. undergoing elective coronary artery bypass graft and/or valve surgery requiring cardiopulmonary bypass
3. English or Spanish-speaking

Exclusion Criteria:

1. severe dementia, neurodegenerative, or psychiatric disease that prevents patient from living independently at baseline
2. emergent surgery
3. inability to perform cognitive testing (i.e. difficulty hearing or inability to speak)
4. contraindications to intranasal administration of medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-jun Jean Hsieh, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine - Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin | Normal Saline
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data besides the amount of patients accrued to each arm are available
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin | Normal Saline | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — Population: The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Age, Continuous [unit: years] — The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available Population: The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Sex: Female, Male — Population: The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Cognitive Function
Description: Assessed using a battery of cognitive tests which test the following four domains: 1) executive function, 2) verbal memory, 3) attention and concentration, 4) language. Cognitive testing will be performed at the following time points: baseline (1-2 weeks prior to surgery) and 6 weeks after discharge.
Time Frame: 6-weeks
Population: The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Delirium and Coma Free Days
Description: Assessed using the Richmond Agitation Sedation Scale (RASS) and Confusion Assessment Method-ICU (CAM-ICU)
Time Frame: 7 days
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Association Between Post-operative Delirium and Post-operative Cognitive Decline
Time Frame: 7 days, 6 weeks
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hypoglycemia
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Nasal Irritation
Time Frame: 14 days
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Survival
Time Frame: 30-day, 90-day
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: ICU Length of Stay
Time Frame: 1 to 90 days
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Hospital Length of Stay
Time Frame: 1 to 90 days
Population: as for outcome 1
Arm/Group | Insulin | Normal Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The PI has left the institution. Efforts were made to contact the PI/study team members on several occasions, but were unsuccessful. No study or adverse event data are available
Arm/Group | Insulin | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution. Efforts were made to contact the PI/study team members on several occasions, but were unsuccessful. Besides the amount of patients accrued to each arm/group, no study or adverse event data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes